CLINICAL TRIAL: NCT06086470
Title: A Prospective Single-Center, Open Label, Non-Randomized Study Evaluating the Use of the Qidni/D Hemodialysis System by Subjects With End-Stage Renal Disease
Brief Title: Evaluating the Use of the Qidni/D Hemodialysis System by Subjects With End-Stage Renal Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qidni Labs Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00061120
Record Dates: First submitted 2023-09-28; First posted 2023-10-17 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Kidney Disease, End-Stage
Keywords: Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, non-randomized study. All participants are enrolled into a single group to be treated with the experimental device.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Treatment Arm (Experimental): Patients will receive one treatment of hemodialysis through the Qidni/D Hemodialysis System.
  Interventions: Device: Qidni/D Hemodialysis System

INTERVENTIONS:
Device: Qidni/D Hemodialysis System — Qidni/D is a hemodialysis device for patients with end-stage renal disease.

SUMMARY:
The main goal of this clinical study is to evaluate the safety of the Qidni/D Hemodialysis System in patients with end-stage renal disease. The main question it aims to answer is:

Is the Qidni/D safe for performing hemodialysis?

Participants will be subjected to one treatment of hemodialysis for up to 4 hours with the use of the Qidni/D.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent.
* Subject is at least 18 years and less than 75 years of age.
* Subject has end-stage renal disease adequately treated by maintenance dialysis and has been deemed stable for at least three months by his/her treating nephrologist.
* Subject has a well-functioning and stable vascular access that allows a blood flow of at least 300 ml/min for conventional treatment or 200-250 mL/min for nocturnal hemodialysis treatment.
* Subject understands the nature of the procedures and the requirements of the study protocol.
* Subject is willing and able to comply with the protocol requirements and return to the treatment center for all required treatments and clinical evaluations.
* Subject has no childbearing potential or the Subject affirms they are not pregnant. Subject affirms using contraception measures to prevent potential pregnancies during the study period.

Exclusion Criteria:

* Subject is unable to read English.
* Subject has dementia or lacks capacity for self-care.
* Life expectancy less than 12 months from first study procedure.
* Subject unable to understand or cooperate with the hemodialysis nurse and dialysis care team.
* Subject has a documented history of non-adherence to dialysis therapy that would prevent successful completion of the study.
* Subject has had a recent major cardiovascular adverse event within the last 3 months.
* Subject has a persistent pre-dialysis sitting systolic blood pressure less than 100 mmHg despite medical therapy.
* Subject has ongoing, symptomatic intra-dialytic hypotension requiring medical intervention.
* Subject has an active infection requiring antibiotics within the last 7 days.
* Subject with fluid overload due to intractable ascites secondary to liver cirrhosis.
* Subject is seroreactive for Hepatitis B Surface Antigen.
* Subject has a history of adverse reactions to dialyzer membrane material.
* Subject is participating in another investigative drug or device clinical study related to dialysis which conflicts with the execution of this study.
* Subject is scheduled to receive an organ transplant during the course of the study: paired exchange or living donor.
* Subject has a life-threatening malignancy actively receiving treatment that would prevent successful completion of the study protocol.
* Any other documented condition that the Investigator feels would prevent the Subject from successful inclusion in the study.
* Subject has an active viral infection (eg. COVID-19).
* Subject is on peritoneal dialysis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-07-14 (Estimated); Study Completion 2024-07-14 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events associated with the use of the Qidni/D device | 3 days
  Adverse events will be recorded and adjudicated independently as to the severity and likelihood of association with treatment with the Qidni/D device.

SECONDARY OUTCOMES:
Efficacy of dialysis | 1 day
  Evaluate the adequacy of dialysis achieved with the Qidni/D device by assessing the change of urea between start and end of dialysis, and compare it to subject's dialysis history.
Efficacy of dialysis | 1 day
  Evaluate the effectiveness of the Qidni/D device in terms of its ability to adequately remove waste products from the subject's blood. This is assessed by the incidence of serum potassium within target range (as established by laboratory normal values) at the end of dialysis treatment.
Efficacy of dialysis | 1 day
  Evaluate the adequacy of dialysis achieved with the Qidni/D device by assessing the change of serum creatinine between start and end of dialysis.
Efficacy of dialysis | 1 day
  Evaluate the adequacy of dialysis with respect to middle molecule clearance achieved with the Qidni/D device by assessing the change of serum beta-2 microglobulin between start and end of dialysis.
Efficacy of dialysis | 1 day
  Evaluate the ability of the Qidni/D device to accurately remove fluid from the subject during dialysis by comparing the device specified targeted fluid removal with the mass of the fluid removed in kilograms.
Hemodynamic stability | 1 day
  Incidence of intradialytic hypotension measured by intradialytic blood pressure less than 90 mmHg systolic with associated symptoms (nausea, vomiting, sweating, dizziness, chest pain).
Technical performance of the Qidni/D device | 1 day
  Number of dialysis sessions interrupted or discontinued due to device malfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Margetts, MD, Principal Investigator — McMaster University
Locations (1):
- Qidni Labs, Kitchener, Ontario, Canada